CLINICAL TRIAL: NCT01619774
Title: An Open-Label Phase II Study of the Combination of GSK2118436 and GSK1120212 in Patients With Metastatic Melanoma Which is Refractory or Resistant to BRAF Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0579; NCI-2012-01222 (Registry Identifier: NCI CTRP); RP120505 (Other Grant/Funding Number: Cancer Prevention Research Institute of Texas (CPRiT))
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic melanoma; Refractory or Resistant to BRAF Inhibitor; Advanced melanoma; GSK2118436; GSK1120212
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2118436 + GSK1120212 (Experimental): GSK1120212 2 mg by mouth once a day, and GSK2118436 150 mg by mouth 2 times every day (1 time in the morning and 1 time in the evening, about 12 hours apart).
  Interventions: Drug: GSK2118436; Drug: GSK1120212

INTERVENTIONS:
Drug: GSK2118436 — Starting dose 150 mg by mouth twice a day.
Drug: GSK1120212 — 2 mg by mouth daily.

SUMMARY:
The goal of this clinical research study is to learn if the combination of 2 drugs dabrafenib and trametinib can help to control melanoma that has or has not spread to the brain. The safety of this drug combination will also be studied.

Dabrafenib is designed to block the mutated BRAF protein. This mutation is only found in moles of the skin and in melanoma cells. By blocking the protein, the drug may slow the growth of or kill cancer cells that have the protein.

Trametinib is designed to block certain proteins that cause cancer cells to grow and multiply. This may cause the cancer cells to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take both dabrafenib and trametinib together.

You will take 1 capsule of trametinib by mouth once a day. You will take 2 capsules of dabrafenib by mouth 2 times every day (1 time in the morning and 1 time in the evening, about 12 hours apart - a total of 4 capsules a day). If you experience severe side effects, your doctor or the research team may lower the dose of the drug(s).

You should take the study drugs with about 1 cup (8 ounces) of room-temperature water. You should not eat or drink anything besides water for at least 1 hour before and 2 hours after you take the study drugs.

You will be given a study drug diary to record the times and doses that you take the study drugs. You should bring the diary to each study visit.

Study Visits:

On Day 1 of Cycle 1:

* Your medical history will be recorded, including any symptoms you may be having. (if it was not recorded in the previous 7 days)
* Your weight, vital signs, and performance status will be recorded.
* You will have a physical exam (if one was not performed in the previous 7 days).
* Blood (about 2 teaspoons) will be collected for routine tests (if this was not performed in the previous 7 days).
* You will be asked about any drugs you may be taking, how you are feeling, and if you have had any side effects.
* You will have a blood draw this visit for research purposes.

At some point between Day 4-10 of Cycle 1, you will have the same kind of biopsy that you had at screening. Your doctor and/or the study team will discuss this with you.

On Days 8 of Cycle 1:

* Your weight, vital signs, and performance status will be recorded.
* Blood (about 4 tablespoons) will be drawn for biomarker testing.
* You will be asked about any drugs or herbal supplements that you may be taking.
* You will be asked about any drugs you may be taking, how you are feeling, and if you have had any side effects.

On Day 15 of Cycle 1:

* You will have a physical exam.
* Your weight, vital signs, and performance status will be recorded.
* You will have an ECG.
* Blood (about 2 teaspoons) will be collected for routine tests.
* Blood (about 4 tablespoons) will be drawn for biomarker testing.
* You will be asked about any drugs you may be taking, how you are feeling, and if you have had any side effects.
* If the disease has spread to the brain and your doctor thinks it is needed, you will have an MRI of the brain.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam.
* Your weight, vital signs, and performance status will be recorded.
* Blood (about 2 teaspoons) will be collected for routine tests.
* You will be asked about any drugs you may be taking, how you are feeling, and if you have had any side effects
* Blood (about 4 tablespoons) will be drawn for biomarker testing on day 1 of Cycle 2 and 4. If your disease worsens, blood (about 4 tablespoons) will also be drawn at that time.

Every 8 weeks (2 cycles) from the time of the start of the treatment, you will have an x-ray, a CT scan, an MRI scan, a skin exam, and/or a bone scan to check the status of the disease.

Every 12 weeks, you will have an ECHO performed.

If at any point during the study you have any symptoms or signs of a serious skin, eye, or heart side effect, you may be referred to a dermatologist or an ophthalmologist, or you may have an ECG and ECHO to check your heart's health.

Length of Study:

You may continue taking the study drugs for as long as the study doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, you start having other health problems, or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

You will have an end-of-study visit within 4 weeks after your last dose of study drugs. The following tests and procedures will be performed:

* You will have a physical exam.
* Your weight, vital signs, and performance status will be recorded.
* You will have an ECG.
* Blood (about 2 teaspoons) will be collected for routine tests. You will have an x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI) scan, and/or bone scan to check the status of the disease if you are taken off the study for any other reason than the disease getting worse.
* Blood (about 4 tablespoons) will be drawn for biomarker testing.
* You will have the same kind of mandatory biopsy that you did at screening. You may be allowed to continue receiving the study drugs until the time of this biopsy (up to 2 days) even if the disease is not showing a response to the study drugs. Your doctor and/or the study team will discuss this with you.

Survival Follow-Up:

After you stop taking study drug, you will be followed approximately every 3 months (either clinic visit or contact by phone or letter) for 5 years or until death. If you are called, the call will last about 5 minutes.

This is an investigational study. This is an investigational study. Both trametinib and dabrafenib are FDA approved and commercially available for the treatment of certain types of melanoma. Their use together in this study is investigational.

Up to 45 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Patients must have histologically or cytologically confirmed Stage IV or recurrent or unresectable Stage III melanoma.
3. BRAF mutation-positive melanoma (i.e., V600E, V600K or V600D)
4. For Cohort A, patients must have easily accessible tumor for a mandatory biopsy. This is not required for patients enrolled on Cohort B.
5. Patients must have measurable disease, defined by RECIST 1.1
6. Patients must have tumor lesions which is refractory or resistant to a selective BRAF inhibitor (RO5185426 or GSK2118436).
7. Age >/= 16 years.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
9. Patients must have organ and marrow function as defined below: · absolute neutrophil count >/= 1,500/mcL · platelets >/= 75,000/mcL · total bilirubin </= 1.5 × institutional upper limit of normal: no restriction to serum bilirubin level if Gilbert's syndrome is diagnosed or suspected · AST(SGOT)/ALT(SGPT) </= 2.5 × institutional upper limit of normal, (</= 3x upper limit of normal for AST and ALT for those subjects with liver metastasis) · creatinine </= 1.3 × institutional upper limit of normal OR · creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels above 1.3 X institutional upper limit of normal.
10. Ability to understand and the willingness to sign a written informed consent document.
11. For Cohort B, patients must have at least 1 measureable parenchymal brain metastasis of at least 10 mm in the greatest diameter and no greater than 40 mm diameter. There must be at least one parenchymal brain metastasis that has not received any previous locally-directed treatment (i.e. surgery or radiation), or that has progressed after prior treatment for the brain metastases (i.e. surgery or radiation).
12. Male subjects must agree to use contraception, this criterion must be followed from the time of the first dose of study medication until 4 weeks after the last dose of study medication. However, it is advised that contraception be used for a total of 16 weeks following the last dose (based on the lifecycle of sperm).
13. A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use contraception if they wish to continue their HRT during the study. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
14. (cont' from Inclusion #12) • Child-bearing potential and agrees to use one of the contraception methods listed in Section 7.1.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 4 weeks after the last dose of study medication, and must have a negative serum pregnancy test within 14 days prior to the start of dosing. Note: Oral contraceptives are not reliable due to potential drug-drug interaction.

Exclusion Criteria:

1. Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) except a selective RAF inhibitor.
2. Patients must not have previously received a selective BRAF inhibitor (RO5185426, GSK2118436) and a selective MEK inhibitor (AZD6244, GSK1120212) concurrently.
3. Received an investigational anti-cancer drug within four weeks or five half-lives (whichever is shorter) of study drug administration, other than BRAF inhibitor--at least 14 days must have passed between the last dose of the prior investigational anti-cancer drug and the first dose of study drug. However, there is no required washout period for any BRAF inhibitors at least until the baseline biopsy is performed.
4. Current use of a prohibited medication or requires any of these medications during treatment with study drug.
5. Any major surgery, within the last 3 weeks. Radiotherapy, or immunotherapy within the last 2 weeks.
6. Unresolved toxicity greater than NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) v4 Grade 1 from previous anti-cancer therapy except alopecia and peripheral neuropathy, for which </= grade 2 toxicity is allowed to participate.
7. Presence of rheumatoid arthritis.
8. History of retinal vein occlusion or central serous retinopathy, or predisposing factors to retinal vein occlusion or central serous retinopathy (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes).
9. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
10. Brain Metastases a. For cohort A, patients will be excluded if they have brain metastases, unless they have been previously treated brain metastases with surgery or stereotactic radiosurgery and the disease has been confirmed stable (i.e., no increase in lesion size) for at least 4 weeks with MRI scans using contrast prior to Day 1. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs and/or steroids to control symptoms/signs of brain metastases. Patients previously treated with whole brain radiation therapy must have confirmed stable disease for at least 12 weeks prior to starting treatment. However, untreated asymptomatic brain metastasis less than 10 mm will be allowed if no steroid and anti-epileptic drugs are used.
11. 10 (con't) b. For cohort B, patients may not have any evidence of leptomeningeal disease. Use of corticosteroids is permitted as long as the dose of steroids required for symptom control has been stable or decreasing for at least 3 weeks prior to the first dose of study treatment.
12. History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 6 months.
13. Corrected QT interval (QTc) >/= 480 msec (>/= 500 msec for subjects with Bundle Branch Block).
14. Uncontrolled arrhythmias. • Subjects with controlled atrial fibrillation for >1 month prior to study Day 1 are eligible.
15. Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
16. Abnormal cardiac valve morphology (subjects with minimal abnormalities can be entered on study if deemed not clinically significant)
17. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients. NOTE: To date there are no known FDA approved drugs chemically related to GSK2118436 or GSK1120212.
18. Pregnant or lactating female.
19. Unwillingness or inability to follow the procedures required in the protocol.
20. Uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity
21. Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davies, MD, PHD, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chen G, McQuade JL, Panka DJ, Hudgens CW, Amin-Mansour A, Mu XJ, Bahl S, Jane-Valbuena J, Wani KM, Reuben A, Creasy CA, Jiang H, Cooper ZA, Roszik J, Bassett RL Jr, Joon AY, Simpson LM, Mouton RD, Glitza IC, Patel SP, Hwu WJ, Amaria RN, Diab A, Hwu P, Lazar AJ, Wargo JA, Garraway LA, Tetzlaff MT, Sullivan RJ, Kim KB, Davies MA. Clinical, Molecular, and Immune Analysis of Dabrafenib-Trametinib Combination Treatment for BRAF Inhibitor-Refractory Metastatic Melanoma: A Phase 2 Clinical Trial. JAMA Oncol. 2016 Aug 1;2(8):1056-64. doi: 10.1001/jamaoncol.2016.0509. PMID 27124486
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 28, 2012 to October 23, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 28 participants screened, five (5) were not eligible following enrollment thus were excluded prior to treatment assignment.
Period: Overall Study
Arm/Group | GSK2118436 + GSK1120212
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK2118436 + GSK1120212
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 54 [27 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate defined as percentage of subjects with a confirmed complete response (CR) or a partial response (PR) at any time as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Clinical responses will be evaluated using RECIST 1.1 criteria after every 2 cycles (8 weeks).
  Complete Response (CR): Disappearance all lesions; pathological lymph nodes reduction in short axis to <10 mm. Partial Response (PR): >30% decrease in sum diameters of lesions, reference baseline sum diameters. Progressive Disease (PD): >20% increase in sum diameters of lesions, reference smallest sum on study (includes baseline sum if smallest on study); relative increase of 20%, sum must also demonstrate absolute increase of >5 mm; appearance of 1 or > new lesions considered progression). Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD, reference smallest sum diameters while on study.
Time Frame: Evaluation every 8 weeks (2 cycles) up to 12 months
Population: Three of the 23 participants were not evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK2118436 + GSK1120212
Number analyzed (Participants) | 20
Percentage of Participants | 10

2. Primary Outcome: Number of Participants by Response
Description: Clinical responses evaluated using RECIST 1.1 criteria after every 2 cycles (8 weeks). Complete Response (CR): Disappearance all lesions; pathological lymph nodes reduction in short axis to <10 mm. Partial Response (PR): >30% decrease in sum diameters of lesions, reference baseline sum diameters. Progressive Disease (PD): >20% increase in sum diameters of lesions, reference smallest sum on study (includes baseline sum if smallest on study); relative increase of 20%, sum must also demonstrate absolute increase of >5 mm; appearance of 1 or > new lesions considered progression). Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD, reference smallest sum diameters while on study.
Time Frame: Evaluation every 8 weeks (2 cycles) up to 12 months
Measure: Number; unit: participants
Arm/Group | GSK2118436 + GSK1120212
Number analyzed (Participants) | 23
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2
  Progressive Disease (PD) | 7
  Stable Disease (SD) | 11
  Not Evaluable | 3

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Duration of response defined for subjects with a confirmed complete response (CR) or partial response (PR), as time from the first documented evidence of a CR or PR until the first documented disease progression or death due to any cause. Progression free survival (PFS) estimated and summarized using the method of Kaplan and Meier.
Time Frame: Evaluation every 8 weeks (2 cycles) up to 12 months
Population: Three of the 23 participants were not evaluable for response therefore not included PFS analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | GSK2118436 + GSK1120212
Number analyzed (Participants) | 20
weeks | 13 [8 to 16]

ADVERSE EVENTS:
Time Frame: Adverse Event collection from the time of the first protocol-specific intervention, through each 4 week cycle until 30 days after the last dose of drug up to 12 weeks.
Arm/Group | GSK2118436 + GSK1120212
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2118436 + GSK1120212 (N=23)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased ejection fraction (Infections and infestations) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2118436 + GSK1120212 (N=23)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Congenital defect (Congenital, familial and genetic disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Confusion (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Investigations - Other Thromobembolic (Investigations) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2)
Social circumstances - mental health issue (Social circumstances) | 2 (2)
Weight loss (Investigations) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 5 (7)
Infection (Infections and infestations) | 6 (6)
Chills (General disorders) | 7 (10)
Pain in extremity (General disorders) | 7 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Blurred vision (Eye disorders) | 7 (7)
Hot flashes (Reproductive system and breast disorders) | 8 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 9 (15)
Anorexia (Metabolism and nutrition disorders) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Headache (Nervous system disorders) | 9 (15)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 12 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 (12)
Constipation (Gastrointestinal disorders) | 13 (15)
Pain (General disorders) | 13 (17)
Fever (Investigations) | 14 (26)
Hypertension (Vascular disorders) | 14 (21)
Dry mouth (Gastrointestinal disorders) | 15 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (16)
Nausea (Gastrointestinal disorders) | 16 (25)
Fatigue (General disorders) | 19 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes